CLINICAL TRIAL: NCT03164668
Title: Menthol Flavored E-cigarette Use During a Simulated Ban of Menthol Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1609M94682
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual cigs; menthol e-cig then tobacco e-cigs (Other): Participants can continue to smoke their usual cigarettes. For the first month of study they receive menthol flavored e-cigarettes and for the second month they receive tobacco flavored e-cigarettes
  Interventions: Other: menthol flavored e-cigarette; Other: tobacco flavored e-cigarette
- Usual cigs; tobacco e-cig then menthol e-cigs (Other): Participants can continue to smoke their usual cigarettes. For the first month of study they receive tobacco flavored e-cigarettes and for the second month they receive menthol flavored e-cigarettes
  Interventions: Other: menthol flavored e-cigarette; Other: tobacco flavored e-cigarette
- avoid menthol cigs; menthol e-cig then tobacco e-cigs (Other): Participants avoid smoking menthol cigarettes. For the first month of study they receive menthol flavored e-cigarettes and for the second month they receive tobacco flavored e-cigarettes
  Interventions: Other: menthol flavored e-cigarette; Other: tobacco flavored e-cigarette
- avoid menthol cigs; tobacco e-cig then menthol e-cigs (Other): Participants avoid smoking menthol cigarettes. For the first month of study they receive tobacco flavored e-cigarettes and for the second month they receive menthol flavored e-cigarettes
  Interventions: Other: menthol flavored e-cigarette; Other: tobacco flavored e-cigarette

INTERVENTIONS:
Other: menthol flavored e-cigarette — menthol flavored e-cigarette
Other: tobacco flavored e-cigarette — tobacco flavored e-cigarette

SUMMARY:
The purpose of this formative study is to provide preliminary data regarding how the availability of menthol flavored e-cigarettes affects tobacco use behavior in the context of a ban on menthol flavored cigarettes

ELIGIBILITY:
Inclusion Criteria:

* Self identify as African American
* smoke primarily menthol cigarettes
* be between the ages of 18 and 64
* smoke a minimum number of cigarettes per day
* agree to abstain from menthol cigarettes for an 8 week period

Exclusion Criteria:

* current unstable medical / psychiatric condition
* regular use any form of nicotine or tobacco other than cigarettes
* are pregnant or breast feeding

The investigators will evaluate if there are other reasons why someone may not be eligible to participate

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Sciences Institute, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants included as having "started" the study are those who completed the baseline visit
Period: Overall Study
Arm/Group | Avoid Menthol Cigs; Menthol E-cig Then Tobacco E-cigs | Avoid Menthol Cigs; Tobacco E-cig Then Menthol E-cigs | Usual Cigs; Menthol E-cig Then Tobacco E-cigs | Usual Cigs; Tobacco E-cig Then Menthol E-cigs
Started | 11 | 7 | 10 | 9
Completed Week 4 | 11 | 5 | 6 | 6
Completed | 10 | 5 | 6 | 6
Not Completed | 1 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Those who completed the Baseline visit of the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Avoid Menthol Cigs; Menthol E-cig Then Tobacco E-cigs | Avoid Menthol Cigs; Tobacco E-cig Then Menthol E-cigs | Usual Cigs; Menthol E-cig Then Tobacco E-cigs | Usual Cigs; Tobacco E-cig Then Menthol E-cigs | Total
Number analyzed (Participants) | 11 | 7 | 10 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11) | 49 (10) | 48 (8) | 47 (14) | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 3 | 15
  Male | 6 | 4 | 6 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 7 | 10 | 9 | 37
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 7 | 10 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Cigarettes Smoked Per Day
Description: Number of cigarettes smoked per day as self-reported on tobacco diary
Time Frame: 1 month
Population: Participants were randomized to either continue to smoke their usual cigarettes or to avoid menthol cigarettes. Within each group, participants received, in random order, one month of menthol flavored e-cigarettes and one month of tobacco flavored e-cigarettes. The overall number of participants entered for each outcome therefore represents the total number from both relevant randomization conditions (see Participant flow for details) in whom at least 1 week of data was provided.
Measure: Number; unit: model estimated cigarettes per day
Groups:
- Avoid Menthol Cigarettes; Menthol E-cigarettes: Participants avoided smoking menthol cigarettes and received menthol flavored e-cigarettes
- Avoid Menthol Cigarettes; Tobacco E-cigarettes: Participants avoided smoking menthol cigarettes and received tobacco flavored e-cigarettes
- Can Continue Smoking Usual Cigarettes; Menthol E-cigarettes: Participants could continue to smoke their usual cigarettes and received menthol flavored e-cigarettes
- Can Continue Smoking Usual Cigarettes; Tobacco E-cigarettes: Participants could continue to smoke their usual cigarettes and received tobacco flavored e-cigarettes
Arm/Group | Avoid Menthol Cigarettes; Menthol E-cigarettes | Avoid Menthol Cigarettes; Tobacco E-cigarettes | Can Continue Smoking Usual Cigarettes; Menthol E-cigarettes | Can Continue Smoking Usual Cigarettes; Tobacco E-cigarettes
Number analyzed (Participants) | 16 | 17 | 13 | 13
model estimated cigarettes per day | 2.2 | 1.8 | 6.0 | 7.1
Statistical Analysis 1: Comparison: Avoid Menthol Cigarettes; Menthol E-cigarettes vs Avoid Menthol Cigarettes; Tobacco E-cigarettes vs Can Continue Smoking Usual Cigarettes; Menthol E-cigarettes vs Can Continue Smoking Usual Cigarettes; Tobacco E-cigarettes; Comparison of those assigned to conditions in which menthol cigarettes are avoided relative to conditions in which can continue smoking usual cigarettes; Test type: Superiority; Estimated mean ratio = 0.31, 95% CI 2-sided [0.13 to 0.72] — Baseline adjusted model estimated mean ratio in cigarettes smoked per day of those randomized conditions in which menthol cigarettes are avoided relative to conditions in which participants can continue smoking usual cigarettes
Statistical Analysis 2: Comparison: Avoid Menthol Cigarettes; Menthol E-cigarettes vs Avoid Menthol Cigarettes; Tobacco E-cigarettes vs Can Continue Smoking Usual Cigarettes; Menthol E-cigarettes vs Can Continue Smoking Usual Cigarettes; Tobacco E-cigarettes; Comparison of those assigned to conditions in which they receive tobacco flavored e-cigarettes relative to conditions in which they receive menthol flavored e-cigarettes; Test type: Superiority; Estimated mean ratio = 0.98, 95% CI 2-sided [0.78 to 1.22] — Baseline adjusted model estimated mean ratio in cigarettes smoked per day among those in conditions in which they receive tobacco flavored e-cigarettes relative to conditions in which they receive menthol flavored e-cigarettes

2. Primary Outcome: Number of E-cigarette Puffs Used Per Day
Description: Self-reported number of puffs of e-cigarettes used per day
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: model estimated e-cig puffs per day
Arm/Group | Avoid Menthol Cigarettes; Menthol E-cigarettes | Avoid Menthol Cigarettes; Tobacco E-cigarettes | Can Continue Smoking Usual Cigarettes; Menthol E-cigarettes | Can Continue Smoking Usual Cigarettes; Tobacco E-cigarettes
Number analyzed (Participants) | 16 | 18 | 16 | 15
model estimated e-cig puffs per day | 61.4 | 57 | 25.5 | 14.9
Statistical Analysis 1: Comparison: Avoid Menthol Cigarettes; Menthol E-cigarettes vs Avoid Menthol Cigarettes; Tobacco E-cigarettes vs Can Continue Smoking Usual Cigarettes; Menthol E-cigarettes vs Can Continue Smoking Usual Cigarettes; Tobacco E-cigarettes; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Estimated mean ratio = 3.03, 95% CI 2-sided [1.39 to 6.61] — Model estimated mean ratio in puffs of e-cigarettes used per day among those randomized to conditions in which menthol cigarettes are avoided relative to conditions in which participants can continue smoking usual cigarettes
Statistical Analysis 2: Comparison: Avoid Menthol Cigarettes; Menthol E-cigarettes vs Avoid Menthol Cigarettes; Tobacco E-cigarettes vs Can Continue Smoking Usual Cigarettes; Menthol E-cigarettes vs Can Continue Smoking Usual Cigarettes; Tobacco E-cigarettes; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Estimated mean ratio = 0.74, 95% CI 2-sided [0.59 to 0.92] — Estimated mean ratio of number of puffs of e-cigarettes used per day among those in conditions in which they receive tobacco flavored e-cigarettes relative to conditions in which they receive menthol flavored e-cigarettes

ADVERSE EVENTS:
Time Frame: For the duration of each participant's participation in the specified condition (up to approximately 4 weeks for each participant)
Description: Adverse events rated as possibly, probably or definitely related to being in the study
Groups:
- Avoid Menthol Cigarettes; Receive Menthol E-cigarettes: Participants avoid smoking menthol cigarettes and receive menthol flavored e-cigarettes
- Avoid Menthol Cigarettes; Receive Tobacco E-cigarettes: Participants avoid smoking menthol cigarettes and receive tobacco flavored e-cigarettes
- Usual Cigarettes; Receive Menthol E-cigarettes: Participants can continue to smoke their usual cigarettes and receive menthol flavored e-cigarettes
- Usual Cigarettes; Receive Tobacco E-cigarettes: Participants can continue to smoke their usual cigarettes and receive tobacco flavored e-cigarettes
Arm/Group | Avoid Menthol Cigarettes; Receive Menthol E-cigarettes | Avoid Menthol Cigarettes; Receive Tobacco E-cigarettes | Usual Cigarettes; Receive Menthol E-cigarettes | Usual Cigarettes; Receive Tobacco E-cigarettes
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 1/18 | 1/16 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avoid Menthol Cigarettes; Receive Menthol E-cigarettes (N=16) | Avoid Menthol Cigarettes; Receive Tobacco E-cigarettes (N=18) | Usual Cigarettes; Receive Menthol E-cigarettes (N=16) | Usual Cigarettes; Receive Tobacco E-cigarettes (N=15)
Headache (General disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lightheaded (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT03164668/Prot_SAP_ICF_000.pdf